CLINICAL TRIAL: NCT01041287
Title: Effect of Nebivolol on Oxidative Stress and Endothelial Progenitor Cells in Subjects With Hypertension
Brief Title: Effect of Nebivolol on Oxidative Stress and Endothelial Progenitor Cells
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00013262; BYD-MD-20 (Other: Other)
Record Dates: First submitted 2009-12-29; First posted 2009-12-31 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol/ Metoprolol (Active Comparator): Subjects were randomized to nebivolol for 3 months. They "crossed over" to take 3 months of metoprolol succinate. The initial 5 mg daily dose of nebivolol was titrated to 10 mg daily after 2 weeks if their BP remained >125/80, and subsequently titrated to 20 mg daily after another 2 weeks if the BP remained >125/80. Similarly, the initial 50 mg daily dose of metoprolol succinate was titrated to 100 mg daily after 2 weeks if BP remained >125/80, and further increased to 200 mg after 2 weeks if BP remained >125/80.
  Interventions: Drug: Nebivolol; Drug: Metoprolol succinate
- Metoprolol/Nebivolol (Active Comparator): Subjects were randomized to metoprolol succinate for 3 months. They "crossed over" to take 3 months of nebivolol. The initial 5 mg daily dose of nebivolol was titrated to 10 mg daily after 2 weeks if their BP remained >125/80, and subsequently titrated to 20 mg daily after another 2 weeks if the BP remained >125/80. Similarly, the initial 50 mg daily dose of metoprolol succinate was titrated to 100 mg daily after 2 weeks if BP remained >125/80, and further increased to 200 mg after 2 weeks if BP remained >125/80.
  Interventions: Drug: Nebivolol; Drug: Metoprolol succinate

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 5 mg PO qday for 2 weeks, titrated up to Nebivolol 10 mg PO qday if BP is >125/80 for the 2 more weeks, and then titrated up to Nebivolol 20 mg PO qday if BP is >125/80 for the remaining 8 weeks
  Other Names: Bystolic
Drug: Metoprolol succinate — Metoprolol 50 mg PO qday for 2 weeks, titrated up to Metoprolol 100 mg PO qday if BP is >125/80 for the 2 more weeks, and then titrated up to Metoprolol 200 mg PO qday if BP is >125/80 for the remaining 8 weeks
  Other Names: Toprol XL

SUMMARY:
Hypertension, or high blood pressure, is a common disease that affects many Americans, and can lead to devastating consequences such as heart attack, stroke, and death if not treated. Nebivolol is a medication that has been recently approved by the FDA for the treatment of hypertension. Nebivolol has an unusual profile compared to other medications, in that its effects may be related to release of a substance called nitric oxide. Nitric oxide is released from the cells lining the blood vessels, and nebivolol may stimulate these cells to release more nitric oxide. Our study will investigate whether treatment with nebivolol, as compared to another medication called metoprolol, in hypertensive subjects will be more effective in protecting blood vessels against the harmful effects of high blood pressure. The mechanisms we will investigate include oxidative stress markers and circulating levels of endothelial progenitor cells.

ELIGIBILITY:
Inclusion Criteria:

1. Males or post-menopausal females aged 21-80 years.
2. Hypertensive patients (BP >135/85) will be eligible to participate.
3. Patients on current anti-hypertensive therapy that does not include beta blockade should have BP >135/85.
4. Patients on anti-hypertensive therapy including beta blockade will have their beta blockers discontinued gradually over 2 weeks before enrolment.
5. Concomitant therapy: Patients will be allowed to be on comcomitant therapy with aspirin, statins, thiazide diuretics, calcium antagonists (for treatment of hypertension), clonidine, vasodilators, or angiotensin antagonists. Patients will be on stable medical therapy for at least 2 months before recruitment. Patients with previous treatment with beta adrenergic blockers (metoprolol, propranolol, atenolol, and labetalol) will also be eligible to participate, but will be randomized to the study beta blocker.

Exclusion Criteria:

1. Age < 21 or >80 years
2. Initiation or change in dose of statin or anti-hypertensive therapy within 2 months before the study
3. Premenopausal females with potential for pregnancy
4. Acute infection in previous 2 weeks
5. History of substance abuse
6. Current neoplasm
7. Chronic renal failure [creatinine > 2.5 mg/dL] or liver failure (Liver enzymes >2X normal)
8. Acute coronary syndrome, Class IV heart failure, CVA, coronary intervention within 2 months
9. Known aortic stenosis, hypertrophic cardiomyopathy.
10. Inability to give informed consent
11. Inability to return to Emory for follow-up testing

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Hayek SS, Poole JC, Neuman R, Morris AA, Khayata M, Kavtaradze N, Topel ML, Binongo JG, Li Q, Jones DP, Waller EK, Quyyumi AA. Differential effects of nebivolol and metoprolol on arterial stiffness, circulating progenitor cells, and oxidative stress. J Am Soc Hypertens. 2015 Mar;9(3):206-13. doi: 10.1016/j.jash.2014.12.013. Epub 2014 Dec 31. PMID 25681236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from clinic sites at Emory University Hospital and by advertisements between December 2009 through April 2012.
Pre-assignment Details: There were 96 subjects enrolled. 58 of the subjects were withdrawn prior to group assignment. 39 subjects did not meet eligibility criteria and 19 subjects withdrew.
Groups:
- Nebivolol/ Metoprolol: Subjects were randomized to nebivolol for the first 3 months. Then they "crossed over" to take 3 months of metoprolol succinate. The initial 5 mg daily dose of nebivolol was titrated to 10 mg daily after 2 weeks if their BP remained >125/80, and subsequently titrated to 20 mg daily after another 2 weeks if the BP remained >125/80. Similarly, the initial 50 mg daily dose of metoprolol succinate was titrated to 100 mg daily after 2 weeks if BP remained >125/80, and further increased to 200 mg after 2 weeks if BP remained >125/80.
- Metoprolol/Nebivolol: Subjects were randomized to metoprolol succinate for the first 3 months. Then they "crossed over" to take 3 months of nebivolol. The initial 5 mg daily dose of nebivolol was titrated to 10 mg daily after 2 weeks if their BP remained >125/80, and subsequently titrated to 20 mg daily after another 2 weeks if the BP remained >125/80. Similarly, the initial 50 mg daily dose of metoprolol succinate was titrated to 100 mg daily after 2 weeks if BP remained >125/80, and further increased to 200 mg after 2 weeks if BP remained >125/80.
Period: Treatment Period 1 (3 Months)
Arm/Group | Nebivolol/ Metoprolol | Metoprolol/Nebivolol
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Treatment Period 2 (3 Months)
Arm/Group | Nebivolol/ Metoprolol | Metoprolol/Nebivolol
Started | 19 | 19
Completed | 16 | 14
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: The population analysis for baseline characteristics are from subjects that completed both treatment periods.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol/ Metoprolol | Metoprolol/Nebivolol | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 28
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Pulse Wave Velocity (Measure of Arterial Stiffness)
Description: The pulse wave velocity (PWV) system measured the velocity of the blood pressure waveform between the carotid and femoral arteries using a single-lead electrocardiogram and tonometer to measure the pressure pulse waveform sequentially at the two peripheral artery sites. PWV is calculated as PWV=distance (d)/time (t) and the unit of measure is reported as meters per second (m/s).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Nebivolol/ Metoprolol | Metoprolol/Nebivolol
Number analyzed (Participants) | 16 | 14
meters per second (m/s) | 9.4 (2.6) | 8.9 (1.5)

2. Primary Outcome: Pulse Wave Velocity (Measure of Arterial Stiffness)
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Nebivolol/ Metoprolol | Metoprolol/Nebivolol
Number analyzed (Participants) | 16 | 14
meters per second (m/s) | 8.4 (2.4) | 10.1 (1.4)

3. Primary Outcome: Pulse Wave Velocity (Measure of Arterial Stiffness)
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Nebivolol/ Metoprolol | Metoprolol/Nebivolol
Number analyzed (Participants) | 16 | 16
meters per second (m/s) | 9.1 (2.2) | 9.8 (1.6)

ADVERSE EVENTS:
Description: 58 subjects were withdrawn prior to randomization/group assignment (no intervention occurred), therefore they are not accounted for in the at-risk population for the adverse events.
Arm/Group | Nebivolol/ Metoprolol | Metoprolol/Nebivolol
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol/ Metoprolol (N=19) | Metoprolol/Nebivolol (N=19)
Stroke (Cardiac disorders) | 0 | 2 — Stroke

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes